CLINICAL TRIAL: NCT03116022
Title: Use of Estriol at Distal Third of the Vaginal Wall Relieving Coital Pain in Women After Menopause: a Randomized, Blinded and Controlled Trial
Brief Title: Use of Estriol at Distal Third of Vagina Improving Coital Pain in Post-menopause Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Lucia Alves da Silva Lara, M.D, Ph.D. Gynecology & Obstetrics, Sexual Health., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 62443916.5.0000.5440
Record Dates: First submitted 2017-03-15; First posted 2017-04-14 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Dyspareunia; Menopause; Sexual Dysfunction
Keywords: menopause; sexual dysfunction; coital pain; vagina
MeSH Terms: conditions — Dyspareunia; Sexual Dysfunction, Physiological | interventions — Estriol; Vaginal Creams, Foams, and Jellies

STUDY DESIGN:
Intervention Model Description: we compared three groups: women using estriol in the proximal vagina wall, women using estriol in the distal vagina wall, and women using gel lubricant
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- proximal estriol group (PEG ) (Active Comparator): This arm is composed of women using estriol 1 mg / 1g in the proximal third of vagina every other night
  Interventions: Drug: Estriol
- distal estriol group (DEG) (Experimental): This arm is composed of women using estriol 1 mg / 1g in the distal third of the vagina every other night
  Interventions: Drug: Distal estriol
- Control group (CG) (Placebo Comparator): This arm is composed of women using vaginal gel lubricant base water during intercourse
  Interventions: Drug: Vaginal Gel

INTERVENTIONS:
Drug: Estriol — Women using drug 1 mg / 1g in the proximal third of the vagina every other night for 12 weeks
  Other Names: PEG
  Arms: proximal estriol group (PEG )
Drug: Distal estriol — Women using drug 1 mg / 1g at the distal third of the vagina every other night for 12 weeks
  Other Names: DEG
  Arms: distal estriol group (DEG)
Drug: Vaginal Gel — Women using a base water gel lubricant during intercourse
  Other Names: CG
  Arms: Control group (CG)

SUMMARY:
Hypoestrogenism leads to vaginal wall changes resulting in diminished vaginal lubrication and, consequently, causing pain during intercourse. Topical estrogen therapy (THT) may control this complaint. However, there are limitations on its use, especially in patients with breast cancer and diagnosed endometrial cancer. This randomized clinical trial aims to assess the impact of local estriol therapy in postmenopausal women complaining of coital pain and to assess serum concentrations of estriol in these women after estriol use. One-hundred-thirty-two women aged between 40 and 65 years will be randomized into three groups: Women using estriol 1 mg / 1g at the proximal third of vagina every other night - estriol proximal group (PEG), women in using estriol 1 mg / 1g at the distal third of the vagina every other night - estriol distal group (DEG), gel group (GG) using water-based during intercourse.

DETAILED DESCRIPTION:
Introduction The daily application of estrogen in the vagina can improve the hydrogen potential (pH), vaginal dryness, burning sensation, dyspareunia, and urinary symptoms. Dyspareunia is highly prevalent after menopause as well as in women after gynecological and breast cancer treatment. However, prescription of topical estrogen therapy (THT) to these women is still controversial, and they are allowed to use only moisturizing cream and vaginal lubricants.

Studies have shown increased serum concentrations of estrogens (estradiol and estrone) after intravaginal suppository containing estradiol use. However, a cohort of 13,479 women treated for breast cancer, 271 received topical hormone therapy (THT), and no increased risk for recurrence was shown in this population.

The main blood supplement to the vagina is mainly from vessels that irrigate proximal vaginal wall, a region where possibly the drug uptake is more intense. However, one study showed that the concentration of estradiol is similarly high regardless of whether the drug was applied to the proximal or distal wall of the vagina. Nevertheless, this study has not been replicated yet.

THT promotes an improvement of coital pain when used in the proximal vagina, but a large population of women with clinical conditions such as thrombophilia and breast cancer cannot benefit from this resource. It is not known if the estriol applied in the distal vagina wall can lead to high serum levels of this hormone.

OBJECTIVES This study aims to evaluate the impact of topic estriol therapy applied in distal vagina wall in coital pain, sexual function, and mood after estriol use. To evaluate serum level of this hormone after estriol use.

METHODS Study design This is a prospective, blind, and randomized clinical trial including post-menopausal women complaining of pain during intercourse. The selected women will be randomized into three groups: estriol proximal group (PEG), estriol distal group (DEG), and gel group (GG). Participants and the assistance staff will not be blinded to the intervention.

Sample Size The sample size was based on the estimated Cohen effect size. Assuming an effect size measure of 0.7 (considered large by Cohen) between groups, and considering a power test of 90% and a significance level of 5%, at least 44 subjects in each arm are required for a total of 132 participants.

Randomization Randomization will be conducted in blocks of random sizes to generate the random allocation sequence. Participants will be randomized in 23 blocks and distributed in intervention groups according to their position in each block.

Participants Sexually-active post-menopausal women between 40 to 65 years old complaining of coital pain will be invited to participate in this study. Sexual activity must include penis-vagina penetration.

Hormonal profile evaluation Blood samples will be collected before the intervention to measure basal serum levels of fasting glucose, thyroid-stimulating hormone (TSH), follicle-stimulating hormone (FSH) and serum estriol. These parameters will be applied in the 12th week of intervention. The measurements of FSH, TSH, and estriol will be performed by chemiluminescence with IMMULITE® 2000 device (DPC IMMULITE® 2000 (Diagnostic Products Corporation, Los Angeles, California, United States of America (USA)). For the measurement of estriol free will be used IMMULITE® kit 2000 unconjugated estriol (SIEMENS, USA). The measurement of hormonal status will be held before the intervention (time 1) and at the end of the intervention (12 weeks). Glucose will be determined by automated spectrophotometry using the liquid enzymatic glycemia kit (Wiener Laboratory, 2000, Rosario, Argentina) Sexual function Sexual function will be evaluated with the Female Sexual Function Index (FSFI). It has 19 questions, with 6 subscales that assess desire, arousal, lubrication, orgasm, satisfaction, and pain. Each question is multiple choice and scored from 0 or 1 to 5. For calculation of the total score (range: 2 to 36), the score of each subscale was multiplied by a factor, and the 6 scores were summed. A lower score corresponds to a worse sexual function, and a score below 26.55 indicates sexual dysfunction.

Emotional condition The Hospital Anxiety and Depression Scale (HAD) was used to assess mood. This scale has 14 items and two subscales, with 7 questions regarding anxiety (HAD-A) and 7 regarding depression (HAD-D). There are four responses to each question (score of 0 to 3), and the sum of scores of each subscale provides a total score from 0 to 21. A cut-off score ≥ 9 for anxiety and depression characterizes the mental state of the woman.

All questionnaires will be applied individually by a gynecologist before the intervention (time 1) and at the end of the intervention (12 weeks) when women attend to collect blood samples. Before applying the questionnaires, women will be informed about the content and objectives of the research, and will also be informed about the issue of confidentiality.

Coital pain evaluation Coital pain will be assessed by the Analogic Visual Scale and the McGill Pain Questionnaire, a multi-dimensional tool that consists of 4 groups of constructs divided into 20 subgroups: Sensory-discriminative group (subgroups 1 to 10) relates to traction, heat, twist, among others; the motivational-affective group (subgroups 11 to 15) describes the affective dimension aspects of tension, as well as fear punishment, and neurovegetative responses; the descriptors of the cognitive component evaluation (subgroup 16) allows the patient to express the overall assessment of the painful experience; subgroups 17-20 comprise miscellaneous items. The subject can choose only one alternative for each subgroup, so the greater the number of most marked pain intensity descriptors, wherein the maximum score is 78. This questionnaire will be applied individually by a gynecologist at the beginning and at 12 weeks of intervention.

INTERVENTION For the PEG group, women will receive professional guidance to use an applicator only 3 cm inside the vagina, once at night, each other night, while lying down to sleep, with a woman in the dorsal position inserting the applicator 3 cm through the vaginal introitus. For the DEG group, women will receive professional guidance to use an applicator totally inside the vagina. The application will be recommended once each other night, while lying down to sleep, with a woman in the dorsal position inserting the applicator 10 cm through the vaginal introitus. Lubricant will be acquired by the researcher in commercial form and should be used during sexual intercourse in the vagina introitus prior to penetration of the penis.

Certification of correct use of prescription A researcher will contact the patient by telephone every two weeks to certify the proper use or any adverse symptoms related to the use of medication.

ETHICAL ASPECTS This project was approved by the Institutional Ethics Committee in Research, and all women shall sign the Informed Consent. This project will be guided according to the ethical standards by Resolution 196/96 of the National Health Council on research with the human being.

Statistical analysis Qualitative variables are described considering the absolute and relative frequencies, as quantitative variables are expressed by central position and dispersion measurements. The comparison between the study groups will be performed using the linear regression model of mixed effects; the model residue analysis will be representing through normal graphics. Cohen measure will be used as the size measure, which is expressed by the difference between the mean divided by the standard deviation. The Statistical Analysis System (SAS) will be used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Women with a clinical diagnosis of menopause
* FSH> 40 milli-International unit (mIU/ml)
* Having sex including penetration of penis into vagina
* Pain during penetration
* Active sexual partners
* Stable relationship.

Exclusion Criteria:

* Previous use of steroids in genital area in the last month
* Thromboembolism history
* Renal insufficiency
* Cholestatic jaundice
* Degenerative vulvar pathology
* Breast cancer
* Endometrial cancer
* Vulvar cancer
* Vaginal cancer history
* Prior radiotherapy to the genital region
* Smoking
* Acute urogenital infections
* Vulvovaginitis
* Urinary tract infection
* Genital herpes
* Genital prolapse grades II, III and IV by Baden Walker
* Systemic hormonal therapy in the last three months
* Use of antidepressants drugs
* Diabetes
* Thyroid disorder
* Cognitive restrictions

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Improvement in pain score after estriol use | baseline and 12 weeks
  Number of women with lower score of pain assessed by the McGill Pain Questionnaire

SECONDARY OUTCOMES:
Number of participants with risk for sexual dysfunction after estriol use | baseline and week 12
  Comparison will be made between the total number of subjects with Female Sexual Function Index (FSFI) total score ≤ 26.55 before after estriol use
Number of participants with risk for anxiety after estriol use | baseline and week 12
  Comparison will be made between the total number of subjects with Hospital Anxiety Scale total score ≥ 9 for anxiety after estriol treatment
Number of participants with risk for depression after estriol use | baseline and week 12
  Comparison will be made between the total number of subjects with Hospital Anxiety Scale total score ≥ 9 for anxiety after estriol treatment
Reduction of de degree of coital pain | baseline and week 12
  Number of women with lower degree of pain accessed by the Analogic Visual Scale graded from 0 to 10, with 0 being no pain and 10 being the maximum level of pain
Variation in serum levels of estriol after estriol use | Assessment of serum concentration of estriol at baseline and week 12.
  Number of women with abnormal laboratory values of estriol after estriol use assessed by chemiluminescence
Variation in serum levels of follicle-stimulating hormone after estriol use | Assessment of serum concentration of follicle-stimulating hormone at baseline and week 12.
  Number of women with abnormal laboratory values of follicle-stimulating hormone after estriol use assessed by chemiluminescence
Variation in serum levels of thyroid-stimulating hormone after estriol use | Assessment of serum concentration of thyroid-stimulating hormone at baseline and week 12.
  Number of women with abnormal laboratory values of thyroid-stimulating hormone after estriol use assessed by chemiluminescence
Number of participants with adverse events that are related to estriol use | Assessment of laboratory values at baseline and week 12. Adverse events assessed each 4 weeks from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 48 months.
  Variation in serum levels of estriol, follicle-stimulating hormone, and thyroid-stimulating hormone will be performed by chemiluminescence. Adverse events will be assessed clinically by telephone
Variation in blood glucose after estriol use | Assessed at baseline and on week 12
  Number of women with abnormal laboratory values for blood glucose determined by the glucose oxidase-phenol (GOD-POD) method
Variation in weight after estriol use Weight | Assessed at baseline and on week 12
  Number of women with weight gain after estriol use
Variation in body mass index (BMI) after estriol use | Assessed at baseline and on week 12
  Number of women with modified BMI after estriol use

CONTACTS AND LOCATIONS:
Overall Officials: lucia a Silva Lara, PhD, Principal Investigator — Faculdade de Medicina de Ribeirão Preto - Universidade de Sao Paulo
Locations (1):
- Hospital das Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lovejoy TI, Turk DC, Morasco BJ. Evaluation of the psychometric properties of the revised short-form McGill Pain Questionnaire. J Pain. 2012 Dec;13(12):1250-7. doi: 10.1016/j.jpain.2012.09.011. PMID 23182230
- [Result] Varoli FK, Pedrazzi V. Adapted version of the McGill Pain Questionnaire to Brazilian Portuguese. Braz Dent J. 2006;17(4):328-35. doi: 10.1590/s0103-64402006000400012. PMID 17262148
- [Result] Weisberg E, Ayton R, Darling G, Farrell E, Murkies A, O'Neill S, Kirkegard Y, Fraser IS. Endometrial and vaginal effects of low-dose estradiol delivered by vaginal ring or vaginal tablet. Climacteric. 2005 Mar;8(1):83-92. doi: 10.1080/13697130500087016. PMID 15804736
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Resplande J, Gholami SS, Graziottin TM, Rogers R, Lin CS, Leng W, Lue TF. Long-term effect of ovariectomy and simulated birth trauma on the lower urinary tract of female rats. J Urol. 2002 Jul;168(1):323-30. PMID 12050564
- [Result] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Result] Simon JA, Maamari RV. Ultra-low-dose vaginal estrogen tablets for the treatment of postmenopausal vaginal atrophy. Climacteric. 2013 Aug;16 Suppl 1:37-43. doi: 10.3109/13697137.2013.807606. PMID 23848490
- [Result] Suckling J, Lethaby A, Kennedy R. Local oestrogen for vaginal atrophy in postmenopausal women. Cochrane Database Syst Rev. 2003;(4):CD001500. doi: 10.1002/14651858.CD001500. PMID 14583935
- [Result] Ting AY, Blacklock AD, Smith PG. Estrogen regulates vaginal sensory and autonomic nerve density in the rat. Biol Reprod. 2004 Oct;71(4):1397-404. doi: 10.1095/biolreprod.104.030023. Epub 2004 Jun 9. PMID 15189832
- [Result] Lara LA, Useche B, Ferriani RA, Reis RM, de Sa MF, de Freitas MM, Rosa e Silva JC, Rosa e Silva AC. The effects of hypoestrogenism on the vaginal wall: interference with the normal sexual response. J Sex Med. 2009 Jan;6(1):30-9. doi: 10.1111/j.1743-6109.2008.01052.x. PMID 19170834
- [Derived] Lara LA, Cartagena-Ramos D, Figueiredo JB, Rosa-E-Silva ACJ, Ferriani RA, Martins WP, Fuentealba-Torres M. Hormone therapy for sexual function in perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2023 Aug 24;8(8):CD009672. doi: 10.1002/14651858.CD009672.pub3. PMID 37619252